CLINICAL TRIAL: NCT01283503
Title: A Phase I Study of BKM120, Administered Orally in Adult Japanese Patients With Advanced Solid Tumors
Brief Title: A Study of BKM120 in Adult Japanese Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120X1101
Record Dates: First submitted 2011-01-13; First posted 2011-01-26 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2016-04

CONDITIONS: Advanced Solid Tumor
Keywords: PI3K,; Advanced solid tumor
MeSH Terms: interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BKM120 (Experimental)
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120

SUMMARY:
In this study, BKM120 will be administered to adult patients with advanced solid tumors whose disease has progressed despite standard therapy or for whom no standard therapy exists. The trial will confirm the safety and tolerability and determine the maximum tolerated dose (MTD) of BKM120 in Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed, advanced unresectable solid tumors who have progressed on (or not been able to tolerate) standard therapy or for whom no standard anticancer therapy exists.
2. At least one measurable or non-measurable lesion as defined by RECIST guidelines for solid tumors.
3. Age ≥ 20 years
4. Eastern Cooperative Oncology Group Performance Status (ECOG P.S.) of ≤ 2
5. Life expectancy of ≥ 12 weeks
6. Patients must have the laboratory values

Exclusion Criteria:

1. Patients with a history of primary central nervous system tumors or brain metastases or who have signs/symptoms attribute to brain metastases and have not been assessed with radiologic imaging to rule out the presence of brain metastases
2. Prior treatment with a PI3K inhibitor
3. Patients with any peripheral neuropathy ≥ CTCAE grade 2
4. Patients with unresolved diarrhea ≥ CTCAE grade 2
5. Women of child-bearing potential who are pregnant or breast feeding. Men or women of reproductive potential not to sign informed consent for birth control. Barrier contraceptives must be used throughout the trial and six months after the end of treatment.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
establish Maximum tolerate dose (MTD) | every day up to first 4 weeks

SECONDARY OUTCOMES:
Safety assessed by type, frequency and severity of adverse events | Every week
Efficacy assessed by RECIST | Every 2 months
Establishment of a pharmacokinetic profile by collecting information on parameters including but not limited to Cmax, Tmax, T1/2 and AUC in plasma samples | Every 2 weeks up to first 4 weeks, then every odd cycle
Measurement of biomarkers for PI3K pathway in blood and tissue | First 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Japan (2):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba

REFERENCES:
- See also: Results for CBKM120X1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7943